CLINICAL TRIAL: NCT03861221
Title: The Technical Operations And Standard Clinical Application Protocol of Cone Beam Breast CT in Diagnostic Process of Breast Cancer
Brief Title: The Technical Operations And Standard Clinical Application Protocol of CBBCT in Diagnostic Process of Breast Cancer
Acronym: CBBCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Collaborators: Sun Yat-sen University (Other); Chinese PLA General Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other); Guangxi Medical University (Other); Koning Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CBBCT2018CIH
Record Dates: First submitted 2019-01-23; First posted 2019-03-04 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2018-06

CONDITIONS: The Clinical Application Guide of Conebeam Breast CT

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Conebeam Breast Computed Tomography (Experimental)
  Interventions: Device: CBBCT

INTERVENTIONS:
Device: CBBCT — To compare the differences between various lesions' presentation on CBBCT and on other approaches under diverse breast conditions.

SUMMARY:
This study intends to recruit about 800 volunteers with 400 malignant cases and 400 benign cases (negative results included). The information acquired from those cases mainly includes: image acquirement parameters, physical examination data of patients, scanning positions, radiological images and diagnosis reports of CBBCT, mammography, breast ultrasound, MRI (if any), pathologic reports, follow-up reports and the like. The image quality comprehensive evaluation and multi-observer, multi-case diagnostic comparing experiment will be processed. With the pathologic report as gold standard, diagnostic comparing experiment between CBBCT and mammography, breast ultrasound, MRI will be designed to determine the differences between various lesions' presentation on CBBCT and on other approaches with diverse breast conditions (size, density).

The problems to be solved in this study include:

1. Standardize the scanning positons, equipment parameter settings and other technical essentials based on the comprehensive analysis of image data acquisition, image quality and diverse patients' conditions, so as to guarantee image quality stability.
2. Summarize the breast anatomic features, typical and atypical lesions' characteristics on CBBCT image based on the analysis of 3D-CBBCT data and pathologic results as well as the comparing of CBBCT with other approaches, so as to establish the radiological diagnostic standard of CBBCT.
3. Standardize the application consensus of CBBCT based on the image features, data acquisition process and patients' conditions.

ELIGIBILITY:
Inclusion Criteria:

* Female, older than 35 years. Already have mammography, or other standard exams (ultrasound, MRI, etc). Could participate this trial within 2 weeks after mammography. Have the ability of consent inform.

Exclusion Criteria:

* During pregnancy or lactation period. Patients that may not be capable of prone position, such as patients with scapulohumeral periarthritis, cardiac pacemaker or have recent cardiac surgery.

Lymphoma patients that under therapy. Severe scoliosis.

Min Age: 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 800 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Standardize the routine scanning and application criteria of CBBCT. | Finish data acquisition and analysis, issue the standardized scanning protocol. Estimated duration: 18 months.
  Standardize the scanning positons, equipment parameter settings and other technical essentials based on the comprehensive analysis of image data acquisition, image quality and diverse patients' conditions; summarize the breast anatomic features, typical and atypical lesions' characteristics on CBBCT; standardize the application guidance of CBBCT based on the image features, data acquisition process and patients' conditions.

SECONDARY OUTCOMES:
Summarize the breast anatomic features and lesions' characteristics on CBBCT. | 1) Finish summarizing the anatomic features of breast on CBBCT. Estimated duration: 12 months. 2)Finish summarizing the typical and atypical lesions' characteristics on CBBCT. Estimated duration: 6 months from when anatomic features summary finished.
  Summarize the breast anatomic features, typical and atypical lesions' characteristics on CBBCT image based on the analysis of 3D-CBBCT data and pathologic results as well as the comparing of CBBCT with other approaches, so as to establish the radiological diagnostic standard of CBBCT.

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoxiang Ye, M.D. & Ph.D., Principal Investigator — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Tianjin Medical University Cancer Institute And Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided